CLINICAL TRIAL: NCT05376189
Title: The Effect of Vitamin D Supplementation on Toll-Like Receptor (TLR) 2, 4, and Clinical Outcomes of Spondylitis Tuberculosis
Brief Title: Oral Vitamin D and Toll Like Receptor in Spondylitis Tuberculosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Assitant Lecturer, Hasanuddin University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0204221709
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Spondylitis; Tuberculosis
Keywords: Vitamin D; Spondylitis Tuberculosis; Clinical Improvement; Toll-Like Receptor
MeSH Terms: conditions — Spondylitis; Tuberculosis | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: This study involves three arms intervention consists of one control group with standardized tuberculosis treatment, and two intervention groups with different level of vitamin D supplementation;
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be masked from the intervention by giving a similar vitamin D preparation in each group. Investigator, Care Provider, and Outcome Assessor are blinded from allocation and only the Allocator knows the participants assigned groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): This group will be given standardized tuberculosis drug with 400 IU of oral Vitamin D3
  Interventions: Dietary Supplement: 400 IU; Drug: Fixed Drug Combination
- Moderate Dose (Experimental): This group will be given standardized tuberculosis drug with 5000 IU of oral Vitamin D3
  Interventions: Dietary Supplement: 5000 IU; Drug: Fixed Drug Combination
- High Dose (Experimental): This group will be given standardized tuberculosis drug with 10000 IU of oral Vitamin D3
  Interventions: Dietary Supplement: 10000 IU; Drug: Fixed Drug Combination

INTERVENTIONS:
Dietary Supplement: 400 IU — An Oral Vitamin D3 400 IU will be given once daily for a total of 8 weeks
  Other Names: Low Dose Vitamin D3
  Arms: Control Group
Dietary Supplement: 5000 IU — An Oral Vitamin D3 5000 IU will be given once daily for a total of 8 weeks
  Other Names: Moderate Dose Vitamin D3
  Arms: Moderate Dose
Dietary Supplement: 10000 IU — An Oral Vitamin D3 10000 IU will be given once daily for a total of 8 weeks
  Other Names: High Dose Vitamin D3
  Arms: High Dose
Drug: Fixed Drug Combination — Standard Tuberculosis Regimen in a form of Fixed Drug Combination (FDC) given for Spondylitis Tuberculosis.
  Other Names: Tuberculosis Regimen

SUMMARY:
Background :

The toll-like receptor is an essential receptor that stimulates the innate immunity response. In tuberculosis, toll-like receptors, particularly the TLR-2, and TLR-4 are crucial in recognizing various ligands with a lipoprotein structure in the bacilli. Vitamin D deficiency leads to lower expression of these receptors, Hence the immune response against Mycobacterium tuberculosis will be altered. Various studies addressed the importance of vitamin D supplementation in pulmonary tuberculosis but the effect of vitamin D in extrapulmonary tuberculosis, particularly spondylitis tuberculosis is not sufficiently identified.

Objectives:

To assess the effect of oral vitamin D supplementation on the expression of TLR-2, TLR-4, and clinical outcomes in spondylitis tuberculosis patients.

Methodology:

This study proposes a randomized clinical trial of oral vitamin D supplementation in spondylitis tuberculosis patients. Multiple arms will be established with different doses and control groups. The outcome of interest includes the clinical outcomes, the expression of TLR-2, and TLR 4

Hypothesis :

It is assumed that oral supplementation of Vitamin D will increase the activation of Toll-Like Receptors and improves the clinical condition of Spondylitis Tuberculosis patients

DETAILED DESCRIPTION:
Target population:

Patients with spondylitis tuberculosis without the involvement of lung and other extrapulmonary infection

Design:

Randomized Clinical Trial with 3 arms

Primary Intervention:

Standardized Tuberculosis treatment with oral Vitamin D3 Supplementation daily for 8 weeks

Outcome:

1. Toll-Like Receptors (TLR) 2 and 4 levels from the blood sample, measured using Enzyme-linked Immunoassay (ELISA).
2. Clinical Evaluation with Visual Analogue Scale (VAS) and Oswestry Disability Index (ODI).

The outcomes will be measured three times at 4-week intervals (baseline, week 4, and week 8)

Sample Size and Recruitment Participants will be recruited from hospitals and allocated by simple randomization

Biological Sample and consent

1. Participants are aware that clinical data collection and biological samples will be obtained by researchers. This is mentioned in informed consent prior to study recruitment
2. Blood sample will be obtained in a standardized phlebotomy procedure and will not be retained after the study is finish.

Hypothesis Sample Size Calculation:

The trial will be designed to compare 2 experimental treatments to a shared control arm.

The sample size was estimated based on the mathematical calculation by a study below Grayling, M.J et al

With the assumption of :

1. K=2 experimental treatments will be included in the trial.
2. A significance level of α=0.05 will be used, in combination with no multiple comparison correction.
3. The event rate in the control arm will be assumed to be: λ0=5.
4. The marginal power for each null hypothesis will be controlled to level 1-β=0.8 under each of their respective least favorable configurations.
5. The interesting and uninteresting treatment effects will be δ1=2.5 and δ0=0 respectively.
6. The target allocation to each of the experimental arms will be the same as the control arm.
7. The sample size in each arm will not be required to be an integer.

Hence total sample should be 37 participants

Proposed Statistical Analysis

1. Descriptive Statistics
2. Bivariate Analysis
3. The study will apply intention-to-treat analysis
4. Linear Mixed model to measure the effect of intervention adjusted by fixed and random factors.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as Spondylitis Tuberculosis (Clinically and Laboratory confirmed)
2. Level of Total Vitamin D <50 nmol/L at baseline

Exclusion Criteria:

1. Participants with pulmonary tuberculosis or other extrapulmonary tuberculosis
2. Participants with osteoporosis, malignancy, cardiovascular disease, diabetes mellitus, and autoimmune disease
3. Participants with liver and kidney dysfunction
4. Participants who received Vitamin D prior to enrollment

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
The Oswestry Disability Index | Changes of Score from Baseline to 8 weeks
  This questionnaire assess the impact of back pain to the daily life. This questionnaire contains 10 6-likert scale questions with the score ranging from 0-5 for each questions. The total score ranging from 0-50. The index is calculated as raw score per total score and presented as percentage. Below is the classification and interpretation of the score:
  0% -20%: Minimal disability 21%-40%: Moderate Disability 41%-60%: Severe Disability 61%-80%: Crippling back pain 81%-100%: These patients are either bed-bound or have an exaggeration of their symptoms
The Visual Analogue Scale | Changes of Score from Baseline to 8 weeks
  This scale represent the pain according to a visual score measured using 10-likert scale. Maximum number indicates extreme/intractable pain
Toll-Like Receptor 2 (TLR-2) | Changes of TLR-2 level from Baseline to 8 weeks
  The level of TLR-2 in blood measured using ELISA
Toll-Like Receptor 4 (TLR-2) | Changes of TLR-4 level from Baseline to 8 weeks
  The level of TLR-4 in blood measured using ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Jainal Arifin, MD, Principal Investigator — Hasanuddin University; Nasrum Massi, MD. Ph.D, Study Chair — Hasanuddin University; Firdaus Hamid, MD. Ph.D, Principal Investigator — Hasanuddin University; Andi Alfian Zainuddin, MD. Ph.D, Principal Investigator — Hasanuddin University
Locations (1):
- Wahidin Sudirohusodo General Hospital, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
As the data is confidential. The data sharing will be granted by investigator upon request

REFERENCES:
- [Background] Grayling MJ, Wason JM. A web application for the design of multi-arm clinical trials. BMC Cancer. 2020 Jan 31;20(1):80. doi: 10.1186/s12885-020-6525-0. PMID 32005187
- [Background] Tang L, Liu S, Bao YC, Gao RX, Han CF, Sun XC, Zhang WL, Feng SQ. Study on the relationship between vitamin D deficiency and susceptibility to spinal tuberculosis. Int J Surg. 2017 Aug;44:99-103. doi: 10.1016/j.ijsu.2017.05.077. Epub 2017 Jun 16. PMID 28629765
- [Background] Panwar A, Garg RK, Malhotra HS, Jain A, Singh AK, Prakash S, Kumar N, Garg R, Mahdi AA, Verma R, Sharma PK. 25-Hydroxy Vitamin D, Vitamin D Receptor and Toll-like Receptor 2 Polymorphisms in Spinal Tuberculosis: A Case-Control Study. Medicine (Baltimore). 2016 Apr;95(17):e3418. doi: 10.1097/MD.0000000000003418. PMID 27124026
- [Background] Ojaimi S, Skinner NA, Strauss BJ, Sundararajan V, Woolley I, Visvanathan K. Vitamin D deficiency impacts on expression of toll-like receptor-2 and cytokine profile: a pilot study. J Transl Med. 2013 Jul 22;11:176. doi: 10.1186/1479-5876-11-176. PMID 23875738
- [Background] Yu, Fang & Cailiang, Shen. (2019). Effect of vitamin D combined with anti-tuberculosis drugs on serum IL-1β, IFN-γ and TH17 cell-associated cytokines for the management of spinal tuberculosis. Tropical Journal of Pharmaceutical Research. 18. 1141-1147. 10.4314/tjpr.v18i5.32.